CLINICAL TRIAL: NCT04376229
Title: Proton Radiation Therapy Registry
Status: Recruiting | Type: Observational
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Other Study IDs: J2008; IRB00228501 (Other: JHM IRB)
Record Dates: First submitted 2020-04-30; First posted 2020-05-06 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Cancer, Therapy-Related
Keywords: proton therapy
MeSH Terms: conditions — Neoplasms, Second Primary | interventions — Registries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients receiving proton radiation therapy: Registry of cancer patients who receive proton radiation therapy to track disease and toxicity outcomes.
  Interventions: Other: Registry

INTERVENTIONS:
Other: Registry — Registry of cancer patients who receive proton radiation therapy

SUMMARY:
The Johns Hopkins Proton Therapy center is establishing a registry to capture the full 3D radiation dosimetry delivered to the patient, baseline clinical data, and disease, toxicity and quality of life outcomes. The goal is to have all patients treated at the proton center to be included in the registry to enable future comparisons of treatment outcomes to assist in understanding which patients can benefit from the use of protons.

DETAILED DESCRIPTION:
Proton based radiation therapy has considerable dosimetric advantages over the standard photon based radiation therapy, with a significantly higher cost. The clinical advantages, however, may not be realized for all patient populations, even with the improved dose distributions. Establishing the clinical efficacy of proton therapy requires years of experience treating patients. The goal is to accelerate the knowledge gain through the use of the registry that allows for detailed information to be captured and is inclusive of every patient treated.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated at the proton center.

Exclusion Criteria:

* Any other than what is supplied in the inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patients with proton therapy
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-04-07 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Research registry of cancer patients receiving proton radiation therapy | 15 years
  This is a clinic based registry of cancer patients' data from participants to be collected over 15 years. The registry will be populated with 3D anatomy and radiation dosimetry from the RayStation treatment planning system used to plan all proton therapy patients. Clinical data will be extracted electronically from the MOSAIQ oncology information system used to manage the radiation therapy treatments. Structured clinical assessments will be routinely captured in the clinical workflow during patient encounters. Patient reported outcomes will be captured with iPad's using the OncoBrowser tools developed in radiotherapy that also interface with MOSAIQ.

CONTACTS AND LOCATIONS:
Overall Officials: Curtiland Deville, MD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Suburban Hospital, Washington D.C., District of Columbia
  - Bayview Hospital, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No